CLINICAL TRIAL: NCT01228149
Title: Investigation of the Efficacy and Safety of Preoperative Intraocular Pressure (IOP) Reduction With Preservative-free COSOPT-S® (Dorzolamide/Timolol, MSD) Eye Drops Versus Oral Acetazolamide and Dexamethasone Eye Drops
Brief Title: COSOPT-S® Treatment Versus Acetazolamide Before Trabeculectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Katrin Lorenz (Other)
Responsible Party: Sponsor-Investigator, Katrin Lorenz, MD, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35131; EUDRA CT 2010-019975-30
Record Dates: First submitted 2010-08-20; First posted 2010-10-26 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-03

CONDITIONS: Glaucoma
Keywords: glaucoma; trabeculectomy; intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diamox/DexaEDO (Active Comparator): Patients receive Diamox (oral acetazolamide) starting 28 days Prior to trabeculectomy. 7 days preoperatively DexaEDO (dexamethasone) eyedrops without preservatives are applied additionally. Patient will undergo trabeculectomy.
  Interventions: Drug: Trabeculectomy with preoperative Diamox/DexaEDO treatment
- Cosopt S (Experimental): Patients receive Cosopt S (dorzolamide/timolol) eye drops starting 28 days before trabeculectomy.
  Interventions: Drug: Trabeculectomy with preoperative Cosopt S treatment

INTERVENTIONS:
Drug: Trabeculectomy with preoperative Diamox/DexaEDO treatment — Filtrating glaucoma surgery, preoperative treatment with Diamox (acetazolamide) 28 day prior surgery. DexaEDO (dexamethasone) 7 days prior surgery
  Other Names: Filtrating glaucoma surgery
  Arms: Diamox/DexaEDO
Drug: Trabeculectomy with preoperative Cosopt S treatment — Filtrating glaucoma surgery, preoperative treatment with Cosopt S (dorzolamide/timolol) 28 day prior surgery.
  Other Names: Filtrating glaucoma surgery
  Arms: Cosopt S

SUMMARY:
The most common cause of post-trabeculectomy filtration failure is postoperative scarring. Long-term preoperative treatment with local antiglaucoma agents containing preservatives has an increased risk of post-operative scarring of the filtration bleb. Therefore many surgeons prepare their patients for planned trabeculectomy by discontinuing local antiglaucoma drugs, controlling IOP with oral acetazolamide, and treating the eye with local steroids.

Preservative-free COSOPT-S® eye drops b.i.d now provide a possibility to reduce IOP preoperatively with the aim of avoiding postoperative excessive scarring and the known adverse effects of oral acetazolamide while achieving comparable IOP reduction and long-term outcomes.

This study will investigate comparability (non-inferiority) of medical benefits of two different IOP lowering pharmaceutical interventions prior to trabeculectomy comparing COSOPT-S® bid to oral acetazolamide plus dexamethasone.

DETAILED DESCRIPTION:
The most common cause of post-trabeculectomy filtration failure is postoperative scarring. Long-term preoperative treatment with local antiglaucoma agents containing preservatives has an increased risk of post-operative scarring of the filtration bleb. Therefore many surgeons prepare their patients for planned trabeculectomy by discontinuing local antiglaucoma drugs, controlling IOP with oral acetazolamide, and treating the eye with local steroids.

Preservative-free COSOPT-S® eye drops b.i.d now provide a possibility to reduce IOP preoperatively with the aim of avoiding postoperative excessive scarring and the known adverse effects of oral acetazolamide while achieving comparable IOP reduction and long-term outcomes.

This study will investigate comparability (non-inferiority) of medical benefits of two different IOP lowering pharmaceutical interventions prior to trabeculectomy comparing COSOPT-S® bid to oral acetazolamide plus dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* Caucasian
* A clinical diagnosis of open angle glaucoma, pseudoexfoliation or pigment dispersion glaucoma, or ocular hypertension in one or both eyes
* Planned trabeculectomy
* Previous treatment with antiglaucoma agents containing preservatives for at least one month
* Best corrected visual acuity of 20/800 or better in the study eye

Exclusion Criteria:

* Secondary glaucoma except pseudoexfoliation glaucoma and pigmentary glaucoma
* Current ocular infection, i.e. conjunctivitis or keratitis
* Any abnormality preventing reliable applanation tonometry
* Intraocular surgery or laser treatment within the past three months
* History of surgery involving the conjunctiva
* History of cataract surgery with sclerocorneal approach
* Subject is allergic to sulfonamides
* Reactive airway disease, including bronchial asthma or a history of bronchial asthma, or severe chronic obstructive pulmonary disease
* Sinus bradycardia, second or third degree atrioventricular block, overt cardiac failure, cardiogenic shock
* Severe renal dysfunction (CrCl < 30 ml/min) or hyperchloraemic acidosis
* Depressed blood levels of sodium and / or potassium
* Marked kidney and liver disease or dysfunction, gout, suprarenal gland failure, hypercalciuria or nephrocalcinosis
* History of hypersensitivity to the investigational medicinal products or to any drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Lorenz, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Clinical Trial Site, Department of Ophthalmology, University Medical Center Johannes Gutenberg University Mainz, Mainz, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Diamox/DexaEDO: Patients receive oral acetazolamide starting 28 days preoperatively. 7 days preoperatively dexamethasone eyedrops without preservatives are applied additionally.
  Trabeculectomy: Filtrating glaucoma surgery, preoperative treatment will be assessed.
- Cosopt S: Patients receive Cosopt S eye drops starting 28 days preoperatively
  Trabeculectomy: Filtrating glaucoma surgery, preoperative treatment will be assessed.
Period: Overall Study
Arm/Group | Diamox/DexaEDO | Cosopt S
Started | 32 | 30
Completed | 27 | 26
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Diamox/DexaEDO: Patients receive Diamox (oral acetazolamide) starting 28 days preoperatively. 7 days preoperatively DexaEDO (dexamethasone) eyedrops without preservatives are applied additionally.
  Trabeculectomy: Filtrating glaucoma surgery, preoperative treatment will be assessed.
- Cosopt S: Patients receive Cosopt S (dorzolamide/timolol) eye drops starting 28 days preoperatively
  Trabeculectomy: Filtrating glaucoma surgery, preoperative treatment will be assessed.
- Total: Total of all reporting groups
Arm/Group | Diamox/DexaEDO | Cosopt S | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 12 | 29
  >=65 years | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.51) | 65.8 (8.82) | 64.98 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 13 | 18 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) (ΔIOP) Three Months After Trabeculectomy in Comparison to the Mean Preoperative IOP
Description: Change in IOP (ΔIOP) three months after trabeculectomy in comparison to the mean preoperative IOP at one day prior surgery
Time Frame: 12 weeks
Population: In total 62 patients were randomized, 30 to COSOPT-S®, 32 to DIAMOX+Dexa edo® (intention-to-treat (ITT) population. Per-protocol (PP) population (treated >8 days and did not take any medication that interfered with the study): n=58 patients: 27 p. in COSOPT-S®, 31 p. in DIAMOX+Dexa edo®. Analysis population: patients who completed the study n=53
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Diamox/DexaEDO: Patients receive oral Diamox (acetazolamide) starting 28 days preoperatively. 7 days preoperatively DexaEDO (dexamethasone) eyedrops without preservatives are applied additionally.
  Trabeculectomy: Filtrating glaucoma surgery, preoperative treatment will be assessed.
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 27 | 26
mmHg | 8.30 [6.85 to 9.75] | 8.12 [6.67 to 9.58]

2. Secondary Outcome: Number of Needling
Description: number of patients requirering needling
Time Frame: 12 weeks
Population: Patients of the PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 31 | 27
Participants | 0 | 2

3. Secondary Outcome: Number of Necessary 5-Fluorouracil (5FU) Injections
Description: Number of post-operative necessary 5-Fluorouracil (5FU) injections at week 12
Time Frame: 12 weeks
Population: PP Population (n=58)
Measure: Mean (Standard Deviation); unit: number of injections
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 31 | 27
number of injections | 5.14 (2.61) | 5.26 (3.13)

4. Secondary Outcome: Ocular Hypotension Rate
Description: Ocular hypotension rate (0-5 mmHg of the study eye) indicated by the number of patients with ocular hypertension
Time Frame: 24 weeks
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 31 | 27
Participants | 5 | 3

5. Secondary Outcome: Change in IOP Between Visit 1 and 2
Description: Change in IOP between Visit 1 (Screening visit 16 to 28 day prior trabeculectomy) and Visit 2 (1 day before trabeculectomy). Outcome shows mean of differences and 95% confidence intervall.
Time Frame: 28 days
Population: PP Population
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 31 | 27
mmHg | 8.19 [5.77 to 10.61] | 1.88 [-0.59 to 4.34]

6. Secondary Outcome: Filtration Bleb Classification
Description: Filtration bleb classification (Grehn) in both Groups 1 week, 4 weeks, 12 weeks and 24 week after surgery.
  For classification the following criteria were evaluated and scored as described below:
  * vascularisation (0=None, 1=mild, 2=a few corkscrew vessels)
  * identifiability (0=no borders to sides; 1=demarcation nasally or temporally; 2= demarcation to both sides; 3= encapsulated)
  * Thickness (0= a least 3mm; 1=2mm; 2= 1mm; 3=flat)
  * Microcysts (0=no; 1= yes)
  * Transparency (0= highly transparent; 2=moderate; 2=not transparent)
  * Mobility (0= yes; 1= no)
  * Leakage (0=yes, 1=no)
  For the change in the filtration bleb classification (only thickness at visit 5/week 12 mentioned below) descriptive statistics were presented only.
Time Frame: 24 weeks
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 31 | 27
Participants
  at least 3 mm | 4 | 2
  2 mm | 14 | 17
  1 mm | 5 | 5
  Flat | 3 | 2
  Missing | 5 | 1

7. Secondary Outcome: Change in Quality of Life
Description: Change in quality of life measure by a certified National Eye Institute Visual Functioning Questionnaire containing 25 questions (NEI VFQ-25).Patients tick a score at every question to present their visual functioning (usually from 1-5 or 1-6 in which 1 is best and 6 worse). Every single item/score is transformed to a scale between 0 and 100 (0 best, 100 worse). For the total score, the mean of all transformed scores/items is calculated.
  NEI VFQ 25 Quality of Life Questionnaire composite score at V5 (week 12 after surgery).
  Outcome shows mean of differences and 95% confidence intervall.
Time Frame: 12 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 32 | 30
scores on a scale | 80.71 (11.64) | 79.48 (15.44)

8. Secondary Outcome: Change in Conjunctival Redness
Description: Conjunctival redness (ORA Scale) evaluated from 16 up to 28 days (time window) prior surgery and 1 day prior surgery. The investigator compares patient's study eye with a set of reference photos showing various degrees of redness. Redness was scored on a scale of "none", "mild", "moderate", "severe" and "very severe". Absolute and relative frequencies of visit 1 and 2 were compared descriptively.
Time Frame: 24 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 32 | 30
Participants
  Visit 1: none | 1 | 0
  Visit 1: mild | 13 | 12
  Visit 1: moderate | 13 | 15
  Visit 1: severe | 4 | 3
  Visit 1: very severe | 1 | 0
  Visit 2: number analyzed (Participants) | 27 | 27
  Visit 2: none | 9 | 7
  Visit 2: mild | 15 | 16
  Visit 2: moderate | 2 | 4
  Visit 2: severe | 1 | 0
  Visit 2: very severe | 0 | 0

9. Secondary Outcome: Number of Suture Lyses
Description: Number of suture lyses at visit 5 (week 12 after surgery)
Time Frame: week 12
Population: Intention-to- treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Diamox/DexaEDO | Cosopt S
Number analyzed (Participants) | 32 | 30
Participants
  0 suture lyses | 11 | 10
  1-2 suture lyses | 10 | 12
  3-4 suture lyses | 7 | 5

ADVERSE EVENTS:
Description: Adverse Event data were colleted from patients with at least one documented treatment with study drug.
Arm/Group | Diamox/DexaEDO | Cosopt S
Serious Adverse Events (participants affected / at risk) | 4/31 | 3/28
Other Adverse Events (participants affected / at risk) | 30/31 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diamox/DexaEDO (N=31) | Cosopt S (N=28)
Cardiac disorders (Cardiac disorders) | 1 | 0
Iris incaceration (Eye disorders) | 0 | 1
Iris neovascularisation (Eye disorders) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0
Musculoskeletal and connective tissue (Investigations) | 0 | 1
Osteoarthritis (Investigations) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diamox/DexaEDO (N=31) | Cosopt S (N=28)
Visual acuity reduced (Eye disorders) | 15 | 15
Paraesthesia (Nervous system disorders) | 14 | 0
Headache (Nervous system disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Atrial faibrillation (Cardiac disorders) | 1 | 0
Weight decreased (Investigations) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Anxietry disorder (Psychiatric disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Eye operation complication (Injury, poisoning and procedural complications) | 5 | 4
Corneal epithelial defect (Eye disorders) | 7 | 0
erythema of eyelid (Eye disorders) | 2 | 4
corneal erosion (Eye disorders) | 2 | 3
eyelid oedema (Eye disorders) | 3 | 1
intraocular pressure increased (Investigations) | 4 | 0
corneal defect (Eye disorders) | 2 | 1
conjunctival haemmorrhage (Eye disorders) | 1 | 2
eye irritation (Eye disorders) | 1 | 2
Hyphaema (Eye disorders) | 3 | 0
Blepharitis (Eye disorders) | 0 | 1
Choroidal detachment (Eye disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 6 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Corneal oedema (Eye disorders) | 1 | 0
Foreign body sensation in eye (Eye disorders) | 0 | 1
Iris incaeceration (Eye disorders) | 0 | 2
Iris Neovascularization (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1
Dizziness (Nervous system disorders) | 7 | 2
Dysgeusia (Nervous system disorders) | 10 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Drug intolerance (General disorders) | 0 | 1
Fatigue (General disorders) | 13 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Fungal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes